CLINICAL TRIAL: NCT06303193
Title: Phase I/II Trial of Pacritinib, a Kinase Inhibitor of CSF1R, IRAK1, JAK2, and FLT3, in Adults and Pediatric Participants 12 Years of Age or Older With Myelodysplastic Syndromes or Myelodysplastic/Myeloproliferative Neoplasms
Brief Title: Pacritinib, a Kinase Inhibitor of CSF1R, IRAK1, JAK2, and FLT3, in Adults and Pediatric Participants 12 Years of Age or Older With Myelodysplastic Syndromes or Myelodysplastic/Myeloproliferative Neoplasms
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001554; 001554-C
Record Dates: First submitted 2024-03-08; First posted 2024-03-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-29

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndrome; bone marrow disorder; Myelodysplasia; myeloproliferative disorders; pediatric bone marrow failure; 5q deletion; multi-lineage dysplasia; Clonal Hematopoiesis; Aplastic Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Bone Marrow Diseases; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Anemia, Aplastic | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I - Pediatric (Experimental): Escalating doses of pacritinib (cohort 1)
  Interventions: Drug: pacritinib
- 2/Phase II - Adult (Experimental): Low-risk cohort (cohort 2): Initiated on pacritinib 100 mg BID. After three cycles, pacritinib dose escalated to 200 mg BID, the adult phase II recommended dose, if not in complete remission.High-risk cohort (cohort 3): Initiated on pacritnib 200 mg BID, the adult phase II recommended dose.
  Interventions: Drug: pacritinib

INTERVENTIONS:
Drug: pacritinib — Pacritinib will be administered orally on a continuous basis for 28 day cycles without a rest period between cycles. Dose assigned by dose level/phase.

SUMMARY:
Background:

Myelodysplastic syndrome (MDS) and myelodysplastic/myeloproliferative neoplasm (MDS/MPN) are blood disorders that can cause serious complications in children and adults. MDS and MDS/MPN can also progress to acute myeloid leukemia. Treatments for these disorders are risky and not always effective. Better treatments are needed.

Objective:

To test a study drug (pacritinib) in adults and children with MDS or MDS/MPN.

Eligibility:

Children (aged 12 to 17 years) and adults (aged 18 years and older) with MDS or MDS/MPN.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have tests of their heart function. They may have a bone marrow biopsy: An area over the hip will be numbed; a needle will be inserted to remove a sample of soft tissue from inside the hipbone.

Pacritinib is a capsule taken by mouth. All participants will take the study drug 2 times a day, every day, in 28-day cycles. They will write down the date and time they take each capsule. Doctors will assign varying dosages of the drug to different participants.

Participants will have clinic visits each week during cycle 1; every 2 weeks during cycle 2; and gradually increasing to every 3 months after cycle 13. Treatment will continue for up to 8 years.

Bone marrow biopsies, heart tests, and other tests will be repeated at intervals throughout the study. Participants will also fill out questionnaires about their quality of life, the symptoms of their disease, and other topics.

DETAILED DESCRIPTION:
Background:

-Myelodysplastic syndromes (MDS) are a heterogeneous group of clonal hematopoietic disorders characterized by peripheral cytopenia, ineffective and dysplastic hematopoiesis, and increased risk of progression to acute myeloid leukemia (AML).

-The significant genetic heterogeneity of MDS contributes to the challenges in treatment.

* Targeting the bone marrow microenvironment (BMME) may allow for treatments that bypass the genetic complexity of MDS.
* MDS studies support a role for changes within the BMME and support the emerging concept that interdependency between the MDS clone and diverse cell populations in the BMME contributes to disease pathophysiology.
* CSF1R is a receptor tyrosine kinase involved in myeloid-lineage cell survival, proliferation, and differentiation.
* The presence of CSF1R-expressing cells in the AML BMME has been shown with evidence that these cells support leukemic cells through cytokine secretion, and the ligand for CSF1R, CSF1, has been shown to be increased in peripheral blood and bone marrow of some patients with MDS, together supporting CSF1R inhibition as a plausible therapeutic target in myeloid malignancies.
* IRAK1, an immune modulating kinase, is overexpressed and hyperactivated in patients with MDS, supporting IRAK1 inhibition as a plausible therapeutic target in MDS.
* A small percentage of patients with MDS have activating mutations in JAK2 or FLT3, and in these patients, JAK2 or FLT3 inhibition may allow for direct anti-tumor effect.
* Pacritinib is a multi-kinase inhibitor of CSF1R, IRAK1, JAK2, and FLT3, all of which are of therapeutic interest in MDS as discussed above and has been overall well tolerated in clinical trials and has shown efficacy in the treatment of myelofibrosis.

Objectives:

-Phase I:

* To determine the safety and confirm the recommended phase II dose of pacritinib in participants who are 12-17 years of age with MDS or MDS/MPN (myelodysplastic/myeloproliferative neoplasms).

  -Phase II:
* To determine the efficacy of pacritinib in participants who are >= 18 years of age with MDS or MDS/MPN, as measured by overall response rate, separately by risk-based cohort.

Eligibility:

-Participants with MDS or MDS/MPN, including therapy-related MDS or MDS/MPN, and MDS or MDS/MPN with germline predisposition, as defined according to the 2016 WHO criteria, 2022 WHO criteria, or 2022 International Consensus Classification

* Age 12-17 years for phase I and age >= 18 years for phase II
* Participants >= 18 years of age with higher-risk MDS (HR-MDS) must have resistance to hypomethylating agents as defined as failure to show improvement after at least 4 cycles of treatment (primary resistance) or relapse in participants with initial response to long-term treatment (secondary resistance) OR have intolerance to hypomethylating agents OR have a contraindication to hypomethylating agents
* Participants >= 18 years of age with LR-MDS must be refractory to OR ineligible to receive standard of care therapies (i.e., erythropoietin-stimulating agents, lenalidomide, luspatercept), and present with one of the following characteristics:

  * Severe neutropenia defined by absolute neutrophils count <=0.5x10^9/L without the use of granulocyte colony-stimulating factors
  * Symptomatic anemia defined by hemoglobin 16-week average <10 g/dL and symptoms that may include fatigue, weakness, reduced exercise tolerance, dyspnea on exertion, palpitations, (orthostatic) hypotension, near syncope and restless legs
  * Thrombocytopenia defined as platelets <20x10^9/L or platelets <50x10^9/L and a history of clinically relevant non-major or major bleeding according to the ISTH classification
* Participants 12-17 years of age with MDS: must be relapsed/refractory OR ineligible to receive immunosuppressive therapy and hematopoietic stem cell transplantation

  * Ineligibility to receive hematopoietic stem cell transplantation will include participants who are not anticipated to be candidates to receive transplantation within the next 3 months due to medical comorbidities, lack of appropriate donor, or logistical barriers

to transplant

* Participants 12-17 years of age must weigh >= 35 kg
* Participants with MDS/MPN must be relapsed/refractory (failed a minimum of 1 standard of care therapy) OR ineligible to receive standard of care OR without known life-prolonging therapy options OR have a diagnosis for which no known standard of care exists

Design:

-This study consists of two phases, which will enroll concurrently:

--Phase I: 3 plus 3 dose-escalation of pacritinib in participants 12-17 years of age with two planned dose levels per group: Group 1 = weight 35 kg to < 50 kg [DL1 = 100 mg BID, DL2 = 200 mg BID], Group 2 = weight >= 50 kg [DL1 = alternating days of 100 mg

BID and 200 mg BID, DL2 = 200 mg BID]

--Phase II: activity evaluation of pacritinib in participants >= 18 years of age, separated into two cohorts:

* Low risk cohort: Initiate on pacritinib 100 mg BID, after completion of 3 cycles, participants will undergo dose escalation to 200 mg BID, the adult phase II recommended dose, unless they meet criteria for complete remission, in which case lower dose pacritinib will be continued without escalation
* High risk cohort: Initiate on pacritinib 200 mg BID, the adult phase II recommended dose

  * In all participants, pacritinib will be administered orally on a continuous basis for cycles of 28 days.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed MDS or MDS/MPN, including therapy-related MDS or MDS/MPN, and MDS or MDS/MPN with germline predisposition, by the Department of Laboratory Medicine Hematology Laboratory, CC or by the Laboratory of Pathology, NCI as defined according to the 2016 WHO criteria, 2022 WHO criteria, or 2022 International Consensus Classification
* Age 12-17 years for phase I and age >= 18 years for phase II
* Participants >= 18 years of age with HR-MDS must have resistance to hypomethylating agents as defined as failure to show improvement after at least 4 cycles of treatment (primary resistance) or relapse in participants with initial response to long-term treatment (secondary resistance) OR have intolerance to hypomethylating agents OR have a contraindication to hypomethylating agents
* Participants >= 18 years of age with LR-MDS must be refractory to or ineligible to receive standard of care therapies, i.e. erythropoietin-stimulating agents, lenalidomide, luspatercept, and present with one of the following characteristics:

  * Severe neutropenia defined by absolute neutrophils count <=0.5(SqrRoot) 10^9/L without the use of granulocyte colony-stimulating factors
  * Symptomatic anemia defined by hemoglobin 16-week average <10 g/dL and symptoms that may include fatigue, weakness, reduced exercise tolerance, dyspnea on exertion, palpitations, (orthostatic) hypotension, near syncope and restless legs
  * Thrombocytopenia defined as platelets <20(SqrRoot) 10^9/L or platelets <50(SqrRoot) 10^9/L and a history of clinically relevant non-major or major bleeding according to the ISTH classification
* Participants 12-17 years of age with MDS must be relapsed/refractory OR ineligible to receive immunosuppressive therapy and hematopoietic stem cell transplantation

  --Ineligibility to receive hematopoietic stem cell transplantation will include participants who are not anticipated to be candidates to receive transplantation within the next 3 months due to medical comorbidities, lack of appropriate donor, or logistical barriers to transplant
* Participants with MDS/MPN must be relapsed/refractory (failed a minimum of 1 standard of care therapy) OR ineligible to receive standard of care OR without known life-prolonging therapy options OR have a diagnosis for which no known standard of care exists
* Participants 12-17 years of age must weigh >= 35 kg
* If any of the prior therapies noted below were given to the participant, they must have been completed within the following timeframes:

  * 7 days from last dose of short-acting myeloid growth factors (i.e., filgrastim) and >= 14 days for long-acting (i.e., pegfilgrastim)
  * 14 days from last dose of short-acting thrombopoietic growth factors (i.e.,eltrombopag) and >= 28 days for long-acting (i.e., romiplostim)
  * 14 days or 5 pharmacokinetic half-lives from biological therapy agent
  * 21 days from myelosuppressive chemotherapy
  * 28 days from last dose of immunosuppressive therapy (e.g., ATG, cyclosporine, steroids greater than physiologic replacement)
  * 28 days from last dose of lenalidomide
  * 28 days from last dose of venetoclax
  * 28 days from any other investigational agent
  * 42 days from last dose of erythropoiesis stimulating agents
  * 56 days from last dose of luspatercept
  * 100 days from stem cell transplant with no evidence of active graft vs. host disease in participants who relapsed following transplant
  * 150 days from total body irradiation
* Performance status:

  * For participants >= 16 years of age, ECOG performance status < 2 (Karnofsky >= 60%)
  * For participants < 16 years of age, Lansky >= 60%
* Participants must have adequate organ function as defined below:

  * Total bilirubin: <= 1.5 X institutional upper limit of normal OR <= 3 x institutional upper limit of normal in participants with Gilbert s syndrome
  * AST(SGOT)/ALT(SGPT): <= 2.5 X institutional upper limit of normal
  * Creatinine clearance: >= 50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
  * PT and PTT: <= 1.5 X institutional upper limit of normal, except in the setting of PTT elevation due to lupus anticoagulant, in which case these participants would be exempt from meeting this inclusion criterion
* Individuals of child-bearing potential (IOCBP) and individuals able to father a child with a partner able to become pregnant must agree to use one (1) highly effective form of contraception (e.g., intrauterine device [IUD], surgical) or two (2) effective forms of contraception (e.g., barrier method) while on study drug and for 30 days after the last dose of study drug
* Nursing participants must discontinue breastfeeding and/or not begin breastfeeding until 2 weeks after the last dose of study drug
* Ability of participant or parent/guardian (for participants 12-17 only) to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Participants with platelet transfusion-refractory thrombocytopenia, with inability to keep platelet threshold above 10 K/mcL with transfusions
* Participants with evidence of ongoing hemorrhage, active signs/symptoms of bleeding, or history of severe (grade >= 3) unprovoked bleeding complications in the one year prior to enrollment, or any unprovoked grade 2 bleeding complications in the 3 months prior

to enrollment

* Use of anti-platelet or anticoagulant medication other than low-dose aspirin (100 mg daily or less) in the 14 days prior to enrollment, or any ongoing requirement for these medications
* Participants who are unwilling to accept blood transfusions
* Participants with ANC < 500 cells/mcL AND hospitalization for a fungal infection in the 12 months prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pacritinib
* Concomitant administration with sensitive substrates/narrow therapeutic index drugs of CYP3A4, CYP1A2, P-gp BCRP, and OCT1 should be avoided. Concurrent use of strong inhibitors and inducers of CYP3A4 are not allowed. Prior use is allowed as long as medication is stopped two weeks prior to study drug initiation. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Concomitant administration of medications with significant potential to cause QTc prolongation.
* Participants with the following cardiac conditions at screening:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac dysrhythmias
  * QTc(F) prolongation >450 ms, or other factors that increase the risk for QT prolongation (i.e., heart failure, or a history of long QT interval syndrome)
* Grade >= 3 cardiac complication in the 6 months prior to enrollment
* Left ventricular ejection fraction <= 50% by transthoracic echocardiogram (TTE) at screening
* Participants with any active, uncontrolled viral, bacterial, or fungal infection, including active HIV-1, Hepatitis B (HBV) and/or Hepatitis C (HCV) infection (positive HBV or HCV viral load in the setting of positive HBV core antibody or surface antibody or HCV antibody); history of HIV, HBV, or HCV is allowed if there is no uncontrolled viral infection
* Pregnancy
* Presence of another known cause of cytopenia or dysplastic marrow that is untreated and may limit interpretation of results
* Uncontrolled intercurrent illness or any significant disease, evaluated by history, physical exam and chemistries or social situations that may limit interpretation of results, limit compliance with study requirements, or that could increase risk to the participant

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of pacritinib in participants 12-17 years of age | 28 days
  Determined by the number of participants with dose-limiting toxicities (DLTs) reported at each dose level studied
Efficacy as measured by Objective Response Rate (ORR) per each risk-based cohort | After every cycle (C4D1, C7D1, C10D1, C16D1) and yearly after
  Clinical responses evaluated by CBC and bone marrow biopsy/aspirate reported separately by cohort, with a separate 95% confidence interval for each cohort

SECONDARY OUTCOMES:
Pharmacokinetic (PK) properties of pacritinib | 28 days
  AUC, half-life, and steady state concentration of pactritinib evaluated separately by dose level using descriptive statistics
Extended safety of pacritinib | Day 1 of study drug through 30 days after the last intervention
  Grades and types of toxicity noted for the agent at each dose level, separately by cohort

CONTACTS AND LOCATIONS:
Overall Officials: Ajoy L Dias, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Kouroukli O, Symeonidis A, Foukas P, Maragkou MK, Kourea EP. Bone Marrow Immune Microenvironment in Myelodysplastic Syndromes. Cancers (Basel). 2022 Nov 17;14(22):5656. doi: 10.3390/cancers14225656. PMID 36428749
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001554-C.html